CLINICAL TRIAL: NCT00725361
Title: A Pilot Study to Evaluate the Efficacy of Ambrisentan in the Treatment and Prevention of Digital Ulcers in Patients With Systemic Sclerosis.
Brief Title: A Study to Evaluate the Efficacy of an Oral Medication in the Treatment and Prevention of Digital Ulcers in Patients With Systemic Sclerosis (Scleroderma).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lorinda S Chung, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-07222008-1265; IRB Protocol # 14409
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: n Ulcer; Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — ambrisentan

ARMS (1):
- Active (Experimental): Ambrisentan
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan

SUMMARY:
This is a research study of an investigational drug called ambrisentan (Letairis) in the treatment and prevention of digital ulcers in patients with systemic sclerosis.

DETAILED DESCRIPTION:
Ambrisentan is an endothelin blocker approved for the treatment of pulmonary arterial hypertension. Patients with systemic sclerosis can have damage to their blood vessels, resulting in increased levels of endothelin in their bloodstream that then causes decreased blood flow to the digits. This can result in very painful digital ulcers. We hope to learn whether blocking the action of endothelin with ambrisentan will be helpful in the treatment and prevention of digital ulcers in patients with systemic sclerosis. This therapy is not approved for the treatment of systemic sclerosis, but this study will help us learn whether ambrisentan is safe and effective in the treatment and prevention of digital ulcers in patients with systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of limited or diffuse systemic sclerosis (SSc) according to American College of Rheumatology or LeRoy criteria
* Age greater than 18 years of age
* At least one digital ulcer located on the volar or lateral surface at or distal to the proximal interphalangeal joints
* At least one new DU that developed within 12 weeks prior to screening
* Vasodilator therapies, including calcium channel blockers, alpha-1-antagonists, ACE-inhibitors, nitroglycerin, and angiotensin receptor blockers, are permitted as long as the doses are stable for 2 weeks prior to screening and throughout the study
* Treatment with omeprazole or other proton pump inhibitors must be stable for 2 weeks prior to screening and throughout the study

Exclusion Criteria:

* Patients with pulmonary arterial hypertension, NYHA Class III or IV
* Patients who are hemodynamically unstable, or have acute renal, cardiac or pulmonary failure
* Concurrent malignancy except non-melanoma skin cancers
* Patients who have required systemic antibiotics for infected digital ulcers within 2 weeks of screening
* Patients receiving phosphodiesterase-5 inhibitors, endothelin receptor antagonists, or prostanoids within 4 weeks of screening
* Patients receiving cyclosporine within 6 weeks of screening
* Patients who have participated in any investigational study within 30 days of screening
* Pregnant or nursing women
* Patients with a history of drug or alcohol abuse within 6 months of screening
* History of hepatitis B, hepatitis C, or HIV infection
* Any medical condition that, in the opinion of the investigator, might interfere with the subject's participation in the study or poses an added risk for the subject
* Inability to comply with study and follow-up procedures
* Transaminase elevation > 3X the upper limit of normal at screening
* Hemoglobin less than 8.5 g/dL
* Platelet count less than 100 X 109/L
* White blood cell count less than 3.0 X 109/L
* Serum creatinine less than 2.0 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorinda S Chung, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ambrisentan: 5 mg orally daily X 4 weeks then 10 mg daily as tolerated
Period: Overall Study
Arm/Group | Ambrisentan
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Active
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 20
Mean number of total baseline digital ulcers [Mean (Standard Deviation); unit: digital ulcers] | 3.1 (2.1)
Mean diameter of baseline digital ulcers [Mean (Standard Deviation); unit: mm] | 3.3 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: New Digital Ulcers (DU) 4 Weeks Prior to Week 24
Description: The number of new digital ulcers (DU) that have developed in the preceding 4 weeks assessed at week 24 from baseline.
Time Frame: 4 weeks prior to week 24
Measure: Mean (Standard Deviation); unit: new digital ulcers
Arm/Group | Active
Number analyzed (Participants) | 16
new digital ulcers | 0.06 (0.68)

2. Secondary Outcome: New DU 4 Weeks Prior to Week 12
Description: The number of new DU that have developed in the preceding 4 weeks assessed at week 12 from baseline.
Time Frame: 4 weeks prior to week 12
Population: At 12 weeks only 1 patient had withdrawn from the study and 19 remained in the study.
Measure: Mean (Standard Deviation); unit: new digital ulcers
Arm/Group | Active
Number analyzed (Participants) | 19
new digital ulcers | -0.26 (1.1)

3. Secondary Outcome: Subjects Experiencing Complete (Total Reepithelialization) Healing of All Baseline DU at Week 12.
Time Frame: 12 weeks
Population: At 12 weeks only 1 patient had withdrawn from the study and 19 remained in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 19
Participants | 7

4. Secondary Outcome: Subjects Experiencing Complete Healing of > 50% of the Number of Baseline DU at Week 12.
Time Frame: 12 weeks
Population: At 12 weeks only 1 patient had withdrawn from the study and 19 remained in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 19
Participants | 12

5. Secondary Outcome: Change in the Scleroderma Health Assessment Questionnaire (SHAQ) at Week 24 Compared With Baseline.
Description: Range is 0-3 with 0 meaning the least amount of disability and 3 the greatest of disability.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active
Number analyzed (Participants) | 16
units on a scale | -0.06 (0.62)

ADVERSE EVENTS:
Time Frame: Screening through week 28 for a total of 32 weeks of data collection.
Arm/Group | Active
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=20)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Raynaud attack (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=20)
Edema (Blood and lymphatic system disorders) | 15
Anemia (Blood and lymphatic system disorders) | 10
Infected digital ulcer (Infections and infestations) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No